CLINICAL TRIAL: NCT04255940
Title: Impact of a Novel Coronavirus (2019-nCoV) Outbreak on Public Anxiety and Cardiovascular Disease Risk in China
Brief Title: 2019-nCoV Outbreak and Cardiovascular Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Pan-Pan Hao, Dr., Qilu Hospital of Shandong University
Other Study IDs: 2019nCoV-CVD
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Cardiovascular Death; Major Adverse Cardiovascular Events

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- After outbreak
- Past 3 months
- Last year

SUMMARY:
Cardiovascular events occurring after 2019-nCoV outbreak in Jinan were prospectively assessed by emergency physicians. We compared those events with events that occurred during the past 3 months and the same months of the last year.

DETAILED DESCRIPTION:
This survey aims to assess whether the public anxiety from a novel coronavirus (2019-nCoV) outbreak increases cardiovascular disease risk in China. Cardiovascular events occurring after 2019-nCoV outbreak in Jinan were prospectively assessed by emergency physicians. We compared those events with events that occurred during the past 3 months and the same months of the last year.

ELIGIBILITY:
Inclusion Criteria:

* Patients visiting emergency department.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients visiting emergency department.
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2020-01-20 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular Death | 3 months

SECONDARY OUTCOMES:
Major Adverse Cardiovascular Events | 3 months
Times From symptom onset to hospital arrival | 3 months
Anxiety | 3 months

CONTACTS AND LOCATIONS:
Locations (12):
- China (12):
  - Affiliated Hospital of Binzhou Medical Universty, Binzhou, Shandong
  - Heze Municipal Hospital, Heze, Shandong
  - Shandong University Qilu Hospital, Jinan, Shandong
  - Jinan Central Hospital, Shandong University, Jinan, Shandong
  - First Hospital Affiliated with Shandong First Medical University, Jinan, Shandong
  - Shandong Provincial Hospital, Shandong University, Jinan, Shandong
  - The Second Hospital of Shandong University, Jinan, Shandong
  - Jining Hospital of Traditional Chinese Medicine, Jining, Shandong
  - Qihe People's Hospital, Qihe, Shandong
  - Affiliated Hospital of Qingdao University Medical College, Qingdao, Shandong
  - Weihai Municipal Hospital, Weihai, Shandong
  - Central Hospital of Zibo, Zibo, Shandong